CLINICAL TRIAL: NCT00449332
Title: Role of Inflammatory and Fibroproliferative Cytokines in the Pathogenesis of Bronchiolitis Obliterans Syndrome-OP in Lung Transplant Recipients.
Brief Title: Early Indicators of Chronic Rejection in Lung Transplant
Acronym: BOS
Status: Terminated | Type: Observational
Why Stopped: PI left University
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 14516A
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Rejection in Lung Transplant; Cytokine Production in Bos Post Lung Transplant
Keywords: Chronic rejection, lung transplant, cytokines, bos
MeSH Terms: conditions — Osteopoikilosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tissues, bal, blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to discover the different patterns of cytokine production in patients who may develop Bronchiolitis Obliterans Syndrome-0p (BOS-0p) which means ongoing rejection. This is an early indicator of chronic rejection in lung transplant recipients. These cytokines can be detected in the bronchoalveolar (lung) and tissue samples of lung transplant recipients.

DETAILED DESCRIPTION:
Lung transplant recipients are routinely followed in clinic every three months after the first year post-transplant. Spirometry with measurement of FEV1, FVC and FEF25-75 are obtained at each visit. In addition, lung transplant recipients undergo surveillance bronchoscopy at one, three, six, nine and twelve months. All bronchoscopy specimens that are obtained for this study will be obtained during bronchoscopies that were scheduled per the physician caring for the patient. An extra 90 cc of sterile solution will be instilled into bronchus and two extra transbronchial biopsies will be performed in addition to the routine bronchoscopic procedure. Routinely, 4-8 transbronchial biopsy samples are obtained from the transplanted lung. Two specimens will be randomly selected for study and the rest will undergo routine histopathologic study. The study biopsies will be set aside and processed. The study visits for this research will occur at the same time as standard of care post transplant visits. We will collect subject's history,demographic of subject's transplant data,donor procurement information, physical exam information, pregnancy tests,blood test and spirometry results from the visits mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipients between the ages of 18 and 65 years old
* All patients must be able to give written informed consent

Exclusion Criteria:

* Lung transplant recipients who are unable to undergo bronchoscopy
* Lung transplant recipients who are unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post lung transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cytokines, chemokines and T cell subsets associated with BOS | 12/2013

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta M Bhorade, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States